CLINICAL TRIAL: NCT05539755
Title: Outcome Indicators of Non-surgical Therapy of Peri-implantitis: a 6-months
Brief Title: Outcome Indicators of Non-surgical Therapy of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Javi Vilarrasa, Clinical Professor, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER-ECL-2020-06
Record Dates: First submitted 2022-09-06; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Peri-Implantitis; Infections
MeSH Terms: conditions — Peri-Implantitis; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-surgical therapy of peri-implantitis (Experimental): Subjects over 18 years old were consecutively included in the study if they present at least one implant in function for more than 1 year diagnosed with peri-implantitis following the case definition of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions (Berglundh et al., 2018).
  Interventions: Procedure: Non surgical debridement of peri-implantitis

INTERVENTIONS:
Procedure: Non surgical debridement of peri-implantitis — The procedure was standardized as follows: the implants' prosthesis was checked for its cleansability, and retrieved when possible. Then, the prosthesis was modified following a previously described elsewhere (de Tapia et al., 2019). After local anaesthesia (articaine 4% and adrenaline 1:100,000), the implant surfaces were cleaned with ultrasonic devices (Newtron P5, Satelec Acteon; Olliergues, France) with the steel alloy H3 dental ultrasonic scaler tip (H3, Satelec Acteon; Olliergues, France), curettage (SyG 7/89 Everdge, Hu-Friedy; Chicago, IL, USA) of the bone defect was performed, and glycine air powder applied submucosally (Air-flow® powder subgingival PERIO, EMS; Nyon, France) with an air-flow piezon device (Air-flow master piezon®, EMS, Nyon; France).
  Oral hygiene instructions were given and metronidazole 500 mg every 8 h for 7 days was prescribed. Patients were scheduled at 3 months for supragingival plaque control and supragingival debridement, if needed.

SUMMARY:
Objectives: To identify patient and implant indicators influencing the non-surgical therapeutic outcomes of peri-implantitis at 6-months follow-up.

Material and methods: This prospective cohort study included patients with at least one implant diagnosed with peri-implantitis according to the 2017 World Workshop. Non-surgical therapy consisted in a mechanical debridement of the peri-implant pockets combined with the metronidazole 500 mg every 8 hours during 7 days. At baseline and at 6 months, clinical and radiographic variables were collected to calculate the success of the therapy. The influence of patient and implant/prosthetic variables on disease resolution were assessed trough simple and multiple logistic regression analysis at patient and implant level using generalized estimation equations models.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years old
* At least one implant in function for more than 1 year diagnosed with peri-implantitis following the case definition of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions (Berglundh et al., 2018).

Exclusion Criteria:

* Previous surgical therapy of peri-implantitis
* Allergy to metronidazole
* Clinical implant mobility
* Pregnancy or lactating females
* Previous non-surgical treatment (i.e., submucosal debridement) of the affected implants at least 12 months before
* Use of systemic antibiotics during the previous 3 months as well as use of systemic antibiotics for endocarditis prophylaxis,
* Systemic diseases, medications, or conditions that may compromise wound healing and influence the outcome of the therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Disease resolution | 6 months
  Probing pocket depth reduction to 5 mm without bleeding on probing (BoP) or <5 mm irrespective to BoP in all implant sites together with lack of progression of peri-implant bone loss

SECONDARY OUTCOMES:
Changes in PPD | From baseline to 6 months
  Measured in mm from the mucosal margin to the base of the peri-implant pocket in 6 sites per tooth
Changes in Bleeding on probing (BoP) | From baseline to 6 months
  Assessed dichotomously (yes/no) in six sites per tooth
Changes in Suppuration on probing (BoP) | From baseline to 6 months
  Assessed dichotomously (yes/no) in six sites per tooth
Changes in soft tissue margin | From baseline to 6 months
  Measured in mm from the mucosal margin to the most apical portion of the crown in 6 sites per tooth
Changes | From baseline to 6 months
  Measured in mm from the mucosal margin to mucogingival line in 6 sites per tooth
Plaque index (PI) | From baseline to 6 months
  Calculated by assigning a binary score to each surface (1 for plaque present, 0 for absent).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No